CLINICAL TRIAL: NCT05243264
Title: Empower@Home: A Feasibility Study of a Novel Internet-based Cognitive Behavioral Therapy Program for Depression Among Homebound Older Adults
Brief Title: Empower@Home: A Feasibility Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Xiaoling Xiang, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00207612
Record Dates: First submitted 2022-01-31; First posted 2022-02-17 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Depression
Keywords: Cognitive Behavioral Therapy; Older Adults; Internet-Based Intervention; Depression; Social Isolation
MeSH Terms: conditions — Depression; Social Isolation

STUDY DESIGN:
Intervention Model Description: The purpose of this research project is to assess the feasibility, acceptability, and preliminary effects of a novel internet-based cognitive behavioral therapy (iCBT) program called Empower@Home. The program is intended to decrease depression in participants by encouraging them to participate in meaningful and enjoyable activities while challenging problematic thinking patterns.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-Based Program (Experimental): Participants will be provided with access to a 10-session online program and will receive supportive remote assistance throughout regarding technical and programmatic issues.
  Interventions: Behavioral: Empower@Home

INTERVENTIONS:
Behavioral: Empower@Home — The intervention is a 10-week course of internet-based cognitive behavioral therapy. During the active intervention phase, participants will receive a weekly check-in call to see how they are doing. The weekly check-in call is intended to be brief and last no more than 10 minutes on average.

SUMMARY:
This is an open pilot feasibility study of a novel internet-based cognitive behavioral therapy program for older adults with elevated depressive symptoms. This study will enroll approximately 15 older adults throughout the state of Michigan to better understand the feasibility of the intervention and to probe preliminary effects. The intervention will take approximately 10 weeks to complete. Participants will have lower levels of depression after completing the intervention than before enrollment. Participants will be able to use the internet-based platform with minimal support.

DETAILED DESCRIPTION:
Depression affects up to 40% of homebound seniors. The purpose of this research project is to assess the feasibility, acceptability, and preliminary effects of a novel internet-based cognitive behavioral therapy (iCBT) program called Empower@Home. Our team developed Empower@Home collaboratively with older adult stakeholders and social service providers. It is the first iCBT program tailored for low-income racially diverse homebound seniors. It has the potential to reduce access barriers to mental health services among this high-need population. Although Empower@Home is based on an evidence-based mental health treatment (i.e., CBT), it is a novel intervention and has not yet been tested with human subjects. This is a pilot study that involves testing the feasibility, acceptability, and preliminary effects of the intervention with a single group of participants in an open trial. No randomization will occur. All eligible participants who consent will receive the intervention. A total of15 older adults will be recruited to participate in this study. All of them will be recruited through referrals from 2 to 3 social service agencies on this list (The Information Center, Region 2 Area Agency on Aging (AAA), Senior Resources, and A & D home care). The intervention involves attending up to 10 pre-recorded online therapy sessions and receiving weekly maintenance calls from trained research assistants for up to 12 weeks. Participants will engage in therapy at their private homes. A comprehensive baseline and post-test will be administered either over the phone or via an online survey, depending on the participants' preference. No in-person interaction between the participants and the research team is anticipated during the active treatment phase unless intervention is warranted for subjects' safety. Quantitative and qualitative data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. ≥60 years
2. have at least mild depressive symptoms, based on PHQ-9 >=5
3. are willing to participate

Exclusion Criteria:

1. Currently receiving CBT or iCBT
2. Probable cognitive impairment based on the Blessed Orientation, Memory, and Concentration scale (score >= 10).
3. They do not speak English
4. have active suicidal ideation (any positive response on the 9th item of PHQ-9)
5. Have a terminal illness or unstable physical health with a high risk of hospitalization within the next 3 months
6. Severe hearing or vision problems that prevent them from using a tablet/computer or viewing online content

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | Change from Baseline PHQ-9 at 12 weeks
  Change in 9 item standardized measures of depressive symptom severity
Modified Treatment Evaluation Inventory | 12 weeks
  11-item Likert scale relating to acceptability of program to participant modified for older adults and the study context

SECONDARY OUTCOMES:
Change in Generalized Anxiety Disorder Assessment-7 (GAD-7) | Change from Baseline at 12 weeks
  Change in 7-item standardized measure for severity of anxiety symptoms
Change in Duke Social Support Index (DSSI)-10 | Change from Baseline at 12 weeks
  Change in 10 item standardized measure for social interaction and satisfaction with social support
Change in PROMISE-SI | Change from Baseline at 12 weeks
  Change in 8 item standardized measure for feelings of loneliness

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoling Xiang, PHD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No